CLINICAL TRIAL: NCT01040091
Title: Cellular Pharmacology of Tenofovir and Emtricitabine for HIV Prophylaxis (Cell Prep)
Brief Title: Evaluation of the Cellular Pharmacology of Tenofovir and Emtricitabine According to HIV Infection Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01 Anderson; 10817 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Racivir; Tenofovir; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-Infected Participants (Active Comparator): HIV-infected participants will receive FTC, TDF, and EFV for 60 days by prescription from their physicians. Participants will receive Truvada (FTC/TDF) and EFV for the first 30 days. After Day 30, participants may switch to the TDF/FTC/EFV co-formulation through Day 60 as directed by their physician.
  Interventions: Drug: Emtricitabine (FTC); Drug: Tenofovir disoproxil fumarate (TDF); Drug: Efavirenz (EFV); Drug: Truvada
- HIV-Uninfected Participants (Active Comparator): HIV-uninfected participants will receive Truvada (FTC/TDF) for 30 days.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Emtricitabine (FTC) — 200 mg once a day
  Arms: HIV-Infected Participants
Drug: Tenofovir disoproxil fumarate (TDF) — 300 mg once a day
  Arms: HIV-Infected Participants
Drug: Efavirenz (EFV) — 600 mg once a day
  Arms: HIV-Infected Participants
Drug: Truvada — 200 mg emtricitabine + 300 mg TDF once a day

SUMMARY:
Tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC) are two antiretroviral medications used for the treatment and prevention of HIV/AIDS. This study will examine how these medications are processed in the body of people who are HIV-infected, as well as in people who are HIV-uninfected.

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate (TDF) and emtricitabine (FTC) are both nucleoside reverse transcriptase inhibitors (NRTIs), a class of medications used for the treatment and prevention of HIV/AIDS. Analyzing how the body interacts with these medications at the cellular level may lead to more effective dosing strategies for both HIV prevention and treatment. This study will examine the pharmacokinetics of TDF and FTC at the cellular level in HIV-infected people (N=20) and HIV-uninfected people (N=20). HIV-infected participants will be allowed to take part in this study only if their doctor already plans to prescribe TDF, FTC, and efavirenz (EFV) for their HIV care, regardless of their participation in this study. HIV-infected participants will receive Truvada (TDF/FTC) and EFV for the first 30 days. After Day 30, participants will continue to receive TDF, FTC, and EFV through Day 60, under the direction of their physician. HIV-infected participants will remain on their therapy throughout the study as part of their HIV care. HIV-uninfected volunteers will receive 30 days of Truvada (TDF/FTC).

The study duration is 60 days. Study visits will occur at baseline and on Days 1, 3, 7, 20, 30, and 60. At most study visits, participants will undergo blood and urine collection for pharmacology studies, a medication history review, and an adverse effects questionnaire. HIV-uninfected participants will also attend two additional study visits at Days 35 and 45 - while off study medication - for blood and urine collection, adverse effects questionnaires, and a medication history review. At varying study visits during the first 30 days, all participants will undergo one rectal biopsy, female participants will undergo one cervical cell and fluid sampling procedure, and male participants will provide one semen sample. In addition to the collections from enrolled participants, study researchers will also analyze previously collected and stored blood samples from participants in the "Chemoprophylaxis for HIV Prevention in Men (iPrEx)" study, which examined the use of TDF and FTC for the prevention of HIV in men who have sex with men (MSM).

ELIGIBILITY:
Inclusion Criteria for HIV-Uninfected Participants:

* Ability to provide informed consent
* Ability to comply with the study procedures

Exclusion Criteria for HIV-Uninfected Participants:

* Positive screening test for HIV infection
* Positive screening test for hepatitis B (HBV) infection
* Pregnant or planning to become pregnant in the 3 months after study entry
* Breastfeeding
* If sexually active and fertile (no tubal ligation or hysterectomy), refusal to use two forms of birth control (e.g., condom and hormonal birth control) during the 60-day study
* Estimated glomerular filtration rate (GFR) less than 60 mL/min/1.73 m^2 by the Modification of Diet in Renal Disease (MDRD) method
* Albuminuria (greater than 30 mg urine albumin per g of urine creatinine)
* Blood donation within 56 days of the screening visit
* Any grade I or higher abnormality in hemoglobin, platelets, serum phosphorous, and lipase on the screening visit; grade I abnormalities in other labs will be evaluated on a case by case basis (using DAIDS criteria)
* Any greater than grade I abnormality in screening laboratory tests (using DAIDS grading criteria)
* Medical history of chronic uncontrolled high blood pressure equal to or above 140/90 mm Hg
* Use of any investigational medication in the 30 days before study entry
* Daily anticoagulant therapy (daily aspirin or non-steroidal anti-inflammatory drugs [NSAIDs] will be allowed if discontinued for 1 week prior to the rectal biopsy)
* Any nephrotoxic concomitant medication (e.g., aminoglycosides, cyclosporine, cidofovir, foscarnet, amphotericin B)
* Active recreational drug or alcohol abuse
* Any concomitant medication (or herbal product) that, in the opinion of the investigators, would interfere with the study outcomes (acceptable medications include acetaminophen, occasional ibuprofen/NSAID, vitamins, and birth control pills)
* History of pathologic bone fractures
* Any chronic or acute medical condition that, in the opinion of the investigator, would interfere with study conditions, such as cancer, heart disease, or diabetes
* Body weight under 110 pounds

Inclusion Criteria for HIV-Infected Participants:

* HIV-infected adults (HIV documented in medical record or by the primary clinician)
* Clinician/participant plan to initiate TDF/FTC/EFV therapy and agree to separate TDF/FTC and EFV prescriptions for the initial 30 days of the study
* Ability to provide informed consent
* Ability to comply with the study procedures

Exclusion Criteria for HIV-Infected Participants:

* Antiretroviral therapy in the preceding 6 months
* Pregnant or planning to become pregnant in the 3 months after study entry
* Breastfeeding
* If sexually active and fertile (no tubal ligation or hysterectomy), refusal to use two forms of birth control (e.g., condom and hormonal birth control) during the 60-day study
* Estimated GFR less than 60 mL/min/1.73 m^2 by the MDRD method
* Albuminuria (greater than 30 mg urine albumin per g of urine creatinine)
* Greater than a grade II abnormality in hemoglobin or platelets. Greater than a grade II abnormality in other clinical chemistry or hematology tests that, in the opinion of the investigators (principal investigator, study coordinator, and study physician) and primary clinician, would preclude participation in the study. DAIDS grading criteria will be used.
* Use of any investigational medication in the 30 days before study entry
* Daily anticoagulant therapy (daily aspirin or NSAIDs will be allowed if discontinued for 1 week prior to the rectal biopsy)
* Any nephrotoxic concomitant medication (e.g., aminoglycosides, cyclosporine, cidofovir, foscarnet, amphotericin B)
* Any concomitant medication (or herbal product) that, in the opinion of the investigators, would interfere with the study outcomes (acceptable medications include acetaminophen, occasional ibuprofen/NSAID, vitamins, and birth control pills)
* Any chronic or acute medical condition that, in the opinion of the investigator, could lead to emergent health complications, or could interfere with the participant's ability to follow study procedures
* Body weight under 110 pounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the first dose tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) area under the concentration-time curve (AUC) in HIV-uninfected adults versus HIV-infected adults | Measured at the time of the first dose
Comparison of average steady-state plasma deoxyguanosine concentrations before therapy and after 30 days of TDF/FTC therapy | Measured through Day 30
Comparison of TFV-DP and FTC-TP in HIV-seroconverters versus matched non-seroconverters from the iPrEx study | Measured throughout the 4-year study
Modeling describing intracellular pharmacokinetics of TFV-DP and FTC-TP in PBMCs so dosing strategies can be tested on the model to identify the optimal dosing that most rapidly achieves and sustains the desired prophylactic threshold for HIV prevention | Measured throughout the 4-year study

SECONDARY OUTCOMES:
Definition of the terminal elimination phase of TFV-DP and FTC-TP in HIV-uninfected adults | Measured from Day 30 to 60
Characterization of TFV-DP and FTC-TP according to cell types: PBMCs, CD4-purified PBMCs (as well as erythrocytes-to include dried blood spot analyses, CD8 cells, B-cells, and monocytes), genital mononuclear cells, and rectal mucosal mononuclear cells | Measured through Day 30
Comparison of TFV-DP and FTC-TP between male and female participants | Measured through Day 30
Characterization of intracellular TFV, tenofovir-monophosphate (TFV-MP), emtricitabine-monophosphate (FTC-MP), and emtricitabine-diphosphate (FTC-DP) | Measured through Day 30
Evaluation of markers of cell activation (HLA-DR and CD38 expression) and the relationship to TFV-DP and FTC-TP concentrations | Measured through Day 30
Effects of TFV-DP and FTC-TP (and plasma EFV) on plasma HIV-RNA and CD4 counts in the HIV-infected participants | Measured through Day 60
Evaluation of relationships between adherence measures collected in iPrEx with TFV-DP and FTC-TP | Measured throughout the 4-year study
Comparison of TFV-DP and FTC-TP between African-American and non-African-American participants | Measured through Day 30
Evaluation of polymorphisms in MRP2 (eg, -24C>T, 1249G>A), MRP4 (eg, 1612C>T, 3463G>A, 3724G>A, 4131T>G), BCRP (eg, 421C>A, 34G>A) and other potentially important enzymes for the study drugs for relationships with pharmacokinetics and pharmacodynamics | Measured throughout the 4-year study
Comparison of Day 30 AUC and overall AUC (AUC over Day 1 to Day 30) TFV-DP and FTC-TP in HIV-uninfected versus HIV-infected participants | Measured through Day 30
HLA-DR / CD38 on T cells will be correlated with changed intracellular and extracellular purine levels in the HIV-uninfected participants to address potential immune-modulation associated with PNP inhibition | Measured throughout the 4-year study
Characterization of the ratios of TFV-DP and FTC-TP to corresponding endogenous deoxyribose nucleotides | Measured throughout the 4-year study
Comparison of TFV-DP and FTC-TP according to iPrEx study sites | Measured throughout the 4-year study

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado CTRC CRS, Aurora, Colorado, United States

REFERENCES:
- [Derived] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401
- [Derived] Chen X, Castillo-Mancilla JR, Seifert SM, McAllister KB, Zheng JH, Bushman LR, MaWhinney S, Anderson PL. Analysis of the Endogenous Deoxynucleoside Triphosphate Pool in HIV-Positive and -Negative Individuals Receiving Tenofovir-Emtricitabine. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5387-92. doi: 10.1128/AAC.01019-16. Print 2016 Sep. PMID 27353267
- [Derived] Castillo-Mancilla JR, Meditz A, Wilson C, Zheng JH, Palmer BE, Lee EJ, Gardner EM, Seifert S, Kerr B, Bushman LR, MaWhinney S, Anderson PL. Reduced immune activation during tenofovir-emtricitabine therapy in HIV-negative individuals. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):495-501. doi: 10.1097/QAI.0000000000000529. PMID 25763783
- See also: Click here for the "Chemoprophylaxis for HIV Prevention in Men (iPrEx)" ClinicalTrials.gov study record. — http://clinicaltrials.gov/ct2/show/NCT00458393